CLINICAL TRIAL: NCT01878890
Title: Phase I Dose Escalation Trial of Efavirenz for Patients With Solid Tumours or Non-Hodgkin Lymphoma in Therapeutic Failure.
Brief Title: Phase I Dose Escalation Trial of Efavirenz in Solid Tumours or Non-Hodgkin Lymphoma in Therapeutic Failure.
Acronym: ESCALE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IB2011-01
Record Dates: First submitted 2012-10-29; First posted 2013-06-17 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Solid Tumors; Non-Hodgkin's Lymphoma
Keywords: Solid tumors (other than pancreas)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — efavirenz

ARMS (4):
- Efavirenz: 600 mg (Experimental): Cohort 1 : Participants received 600 mg of Efavirenz (oral / once a day), until progression or toxicity.
  Interventions: Drug: Efavirenz 600mg
- Efavirenz: 1200 mg (Experimental): Cohort 2 : Participants received 1200 mg of Efavirenz (oral / once a day), until progression or toxicity.
  Interventions: Drug: Efavirenz 1200 mg
- Efavirenz: 1800 mg (Experimental): Cohort 3 : Participants received 1800 mg of Efavirenz (oral / once a day), until progression or toxicity.
  Interventions: Drug: Efavirenz 1800 mg
- Efavirenz: 2200 mg (Experimental): Cohort 4 : Participants received 2200 mg of Efavirenz (oral / once a day), until progression or toxicity.
  Interventions: Drug: Efavirenz 2200 mg

INTERVENTIONS:
Drug: Efavirenz 600mg — Efavirenz 600 mg (oral daily intake)
  Arms: Efavirenz: 600 mg
Drug: Efavirenz 1200 mg — Efavirenz 1200mg (oral daily intake)
  Arms: Efavirenz: 1200 mg
Drug: Efavirenz 1800 mg — Efavirenz 1800mg (oral daily intake)
  Arms: Efavirenz: 1800 mg
Drug: Efavirenz 2200 mg — Efavirenz 2200mg (oral daily intake)
  Arms: Efavirenz: 2200 mg

SUMMARY:
Hypothesis: encouraging results of phase II study FAVE in the treatment of hormonal resistant prostate cancer lead us to continue clinical development of efavirenz. Furthermore, all available pre-clinical and clinical data lead us to conduct a Phase 1 study with efavirenz. Objective of this Phase I is to test doses above 600 mg / day in patients with cancer in order to determine the maximum tolerated dose to improve therapeutic effect.

This study is a single center Phase I trial, conduct with dose escalation scheme of efavirenz by continual reassessment method likehood approach (CRML) on solid tumours (except pancreatic cancer) and non-Hodgkin lymphoma (NHL).

Main objective is to determine the safety profile, and particularly the maximum tolerated dose of efavirenz for the treatment of patients with solid tumors (except pancreatic cancer) or NHL in therapeutic failure.

Secondary objectives are:

* Evaluate efavirenz pharmacokinetics at 2, 4 and 12 weeks;
* Evaluate objective response at 12 weeks;
* Evaluate progression free survival at 6 months;
* Assess biological progression-free survival at 6 months (prostate tumours only).

Primary Endpoint

Safety will be evaluated according to the toxicity scale NCI-CTCAE v4.0. Dose limiting toxicities will be collected during the first 28 days (+ / - 7 days) after first dose of Efavirenz and will be defined as follows:

* Any drug-related toxicity with grade ≥ 3 according to NCI-CTCAE v4.0 (except alopecia, nausea and vomiting, regardless of grade),
* Any drug-related toxicity, regardless of grade, who led a treatment delay> 14 days,
* Score ≥ 19 HAD during treatment. Secondary Criteria
* Solid tumors: response and progression defined by RECIST v1.1 [Eisenhauer EA et al. EJC 2009).
* Non-Hodgkin lymphomas: Response and progression defined according to Cheson criteria [Cheson BD et al. JCO 1999]
* Biological progression (particular case of prostate tumors): defined according to Scher [Scher HI et al. JCO 2008] Statistical Considerations This is a Phase I dose escalation strategy using the method CRML, described by O'Quigley and Shen [O'Quigley et al. Biometrics 1996] and commonly used in Phase I trials in oncology.
* Maximum number of eligible and evaluable subjects is 30.
* Six dose levels are initially defined: 600 mg, 1200 mg, 1800 mg, 2200 mg, 2600 mg, 3000 mg.
* The risk of dose limiting toxicities maximum allowed is 25%.

DETAILED DESCRIPTION:
This is a Phase I dose escalation strategy according to the method described by CRML O'Quigley and Shen [O'Quigley et al. Biometrics 1996] and commonly used in phase I trials in oncology.

Six levels of doses are initially defined: 600 mg, 1200 mg, 1800 mg, 2200 mg, 2600 mg, 3000 mg.

The maximum potential dose-limiting toxicities allowed is 25%.

Dose limiting toxicities will be defined as follows:

* Any drug-related toxicity with grade ≥ 3 according to NCI-CTCAE v4.0 (except alopecia, nausea and vomiting, regardless of grade),
* Any drug-related toxicity, regardless of grade, who led a treatment delay> 14 days,
* Score ≥ 19 HAD during treatment.

ELIGIBILITY:
Inclusion Criteria :

1. Patients with solid tumors (except pancreatic cancer) or non-Hodgkin lymphoma
2. Metastatic disease or locally advanced inoperable tumor, not accessible to standard therapy.
3. Male or female ≥ 18 years and <80 years.
4. Tumor assessable by RECIST v1.1, Scher Cheson 2008 or 99.
5. At least 28 days after completion of prior treatment (radiotherapy, systemic chemotherapy or major surgery).
6. Patient who recovered from any prior toxicity ≤ grade 1.
7. WHO 0-1 in the 7 days before inclusion.
8. Neutrophils ≥ 1500/mm3, Platelets ≥ 100 000/mm3.
9. Total bilirubin and serum creatinine within normal limits (≤ 1.5 ULN), creatinine clearance ≥ 40 ml / min.
10. AST / ALT ≤ 1.5 ULN (≤ 5 ULN if liver metastasis).
11. Normal thyroid function.
12. Normal coagulation: TP ≥ 70%.
13. Life expectancy upper than 3 months.
14. HAD score <13.
15. Negative pregnancy test for women likely to be pregnant within 7 days before inclusion.
16. Effective contraception for the duration of treatment (for both sexes in childbearing or reproductive age): mechanic contraception method should always be used in combination with other contraceptive methods (eg, oral or other hormonal contraceptives). Because of long half-life of efavirenz, it is recommended to use adequate contraceptive measures for 12 weeks after stopping treatment with efavirenz.
17. Informed consent signed and dated by the patient or his legal representative before the establishment of any specific procedure to the study.
18. Clinical examination and laboratory tests made within 7 days before enrollment and start of treatment.
19. Initial assessment and radiological CT / or MRI performed within 30 days before enrollment.
20. Patients potentially compliant with treatment and follow-up study.
21. Ability to swallow capsules or tablets.
22. Patients insured by a social security system.

Exclusion Criteria :

1. Patient with pancreatic cancer.
2. Presence of active or symptomatic cerebral localization (known).
3. History of another cancer except:

   * cancer occurred more than five years and considered in complete remission
   * in situ cervix carcinomas,
   * cutaneous basal cell carcinomas.
4. Current major depressive state (screening by HAD scale total score ≥ 13).
5. Patients with history of depressive disorders, suicide attempts, addiction or other psychiatric disorders.
6. Concomitant use of terfenadine, astemizole, cisapride, midazolam, triazolam, pimozide, bepridil, alkaloids of ergot, voriconazole, mixing St. John's Wort.
7. Patients treated with anti-vitamin K. Treatment with low molecular weight heparin are allowed.
8. Known efavirenz hypersensitivity or to any of its excipients.
9. Severe renal impairment.
10. Severe hepatic impairment.
11. Yellow fever vaccine (yellow fever).
12. Pregnant or lactating.
13. Presence of toxicity> 1 according to the criteria CTCAE V4.0, due to prior cancer therapy.
14. Recurrent diarrhea which can interfere with drug absorption capacity.
15. Patient included in another biomedical research on a drug within 30 days of inclusion.
16. Patient who previously participated in this study.
17. Patient, who for reasons psychological, psychiatric, social, family or geographical could not be treated or monitored regularly by the criteria of the study, patients deprived of liberty or under tutorship.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-09-05 (Actual); Primary Completion 2014-09-16 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guilhem Roubaud, MD, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Efavirenz - 600 mg: Participants received 600 mg of Efavirenz (oral / once a day), until progression or toxicity.
- Efavirenz - 1200 mg: Participants received 1200 mg of Efavirenz (oral / once a day), until progression or toxicity.
- Efavirenz - 1800 mg: Participants received 1800 mg of Efavirenz (oral / once a day), until progression or toxicity.
- Efavirenz - 2200 mg: Participants received 2200 mg of Efavirenz (oral / once a day), until progression or toxicity.
Period: Overall Study
Arm/Group | Efavirenz - 600 mg | Efavirenz - 1200 mg | Efavirenz - 1800 mg | Efavirenz - 2200 mg
Started | 5 | 11 | 4 | 5
Completed | 5 | 10 | 4 | 5
Not Completed | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Efavirenz: 1200 mg: Cohort 2 : Participants received 1200 mg of Efavirenz (oral / once a day), until progression or toxicity.
  Efavirenz 600mg: Efavirenz 1200 mg (oral daily intake)
- Efavirenz: 1800 mg: Cohort 3 : Participants received 1800 mg of Efavirenz (oral / once a day), until progression or toxicity.
  Efavirenz 600mg: Efavirenz 1800 mg (oral daily intake)
- Efavirenz: 2200 mg: Cohort 4 : Participants received 2200 mg of Efavirenz (oral / once a day), until progression or toxicity.
  Efavirenz 600mg: Efavirenz 2200 mg (oral daily intake)
- Total: Total of all reporting groups
Arm/Group | Efavirenz: 600 mg | Efavirenz: 1200 mg | Efavirenz: 1800 mg | Efavirenz: 2200 mg | Total
Number analyzed (Participants) | 5 | 10 | 4 | 5 | 24
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 64.4 [62 to 66.4] | 59.0 [51.5 to 70] | 66.8 [63.1 to 70.4] | 63.4 [62.7 to 67.7] | 62.2 [59.5 to 68.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 1 | 9
  Male | 3 | 7 | 1 | 4 | 15
Region of Enrollment [Number; unit: participants]
  France | 5 | 10 | 4 | 5 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Efavirenz
Description: MTD was determined by testing increasing doses up to 3000 mg (oral daily intake).
  The dose escalation scheme is the continual reassessment method likehood approach (CRML) described by O'Quigley and Shen [O'Quigley et al. Biometrics 1996].
  MTD reflects the highest dose of drug that did not cause a Dose-Limiting Toxicity (DLT) in > 25% of participants.
  A DLT was any drug-related toxicity with grade ≥ 3 according to NCI-CTCAE v4.0 (except alopecia, nausea and vomiting, regardless of grade), any drug-related toxicity, regardless of grade, who led a treatment delay> 14 days, a score ≥ 19 for the Hospital Anxiety And Depression Scale (HAD) during treatment.
Time Frame: Up to 28 days for each dosing cohort
Measure: Number; unit: mg
Groups:
- All Participants: All participants who received at least 1 dose of Efavirenz, either at 600 mg, 1200 mg, 1800 mg, or 2200 mg.
Arm/Group | All Participants
Number analyzed (Participants) | 25
mg | 1200

2. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: A DLT was any drug-related toxicity with grade ≥ 3 according to NCI-CTCAE v4.0 (except alopecia, nausea and vomiting, regardless of grade), any drug-related toxicity, regardless of grade, who led a treatment delay> 14 days, a score ≥ 19 for the Hospital Anxiety And Depression Scale (HAD) during treatment.
Time Frame: Up to 28 days for each dosing cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Efavirenz: 600 mg | Efavirenz: 1200 mg | Efavirenz: 1800 mg | Efavirenz: 2200 mg
Number analyzed (Participants) | 5 | 10 | 4 | 5
Participants | 0 | 3 | 1 | 3

3. Secondary Outcome: 12-week Objective Response Rate
Description: Objective response is defined as complete or partial response (CR, PR) using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Objective reponse rate is calculated as the number of patients with objective reponse divided by the number of alive patients.
Time Frame: up to 3 months after first adminitration of Efavirenz
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 24
Participants | 0

4. Secondary Outcome: 12-week Non-progression Rate
Description: Non progression is defined as complete or partial response (CR, PR) or stable disease (SD), using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Non-progression rate is calculated as the number of alive and progression free patients divided by the number of patients.
Time Frame: Evaluated up to 3 months after first administration of Efavirenz
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 24
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected until death or date of the end of study (6 months after the inclusion of the last patient)
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Arm/Group | Efavirenz: 600 mg | Efavirenz: 1200 mg | Efavirenz: 1800 mg | Efavirenz: 2200 mg
All-Cause Mortality (participants affected / at risk) | 5/5 | 11/11 | 4/4 | 5/5
Serious Adverse Events (participants affected / at risk) | 3/5 | 4/11 | 4/4 | 3/5
Other Adverse Events (participants affected / at risk) | 5/5 | 11/11 | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efavirenz: 600 mg (N=5) | Efavirenz: 1200 mg (N=11) | Efavirenz: 1800 mg (N=4) | Efavirenz: 2200 mg (N=5)
Other (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Other (General disorders) | 0 (0) | 2 (2) | 4 (7) | 2 (3)
other (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Other (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (2)
other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Efavirenz: 600 mg (N=5) | Efavirenz: 1200 mg (N=11) | Efavirenz: 1800 mg (N=4) | Efavirenz: 2200 mg (N=5)
Not collected (Blood and lymphatic system disorders) | 1/1 (1) | 2 (2) | 2 (2) | 0 (0)
Not collected (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Not collected (Gastrointestinal disorders) | 4 (7) | 8 (12) | 3 (4) | 3 (7)
Not collected (General disorders) | 3 (3) | 8 (11) | 4 (7) | 5 (9)
Not collected (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Not collected (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Not collected (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Not collected (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Not collected (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Not collected (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Not collected (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Not collected (Nervous system disorders) | 2 (2) | 5 (6) | 0 (0) | 4 (5)
Not collected (Psychiatric disorders) | 0 (0) | 6 (8) | 2 (3) | 5 (12)
Not collected (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Not collected (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Not collected (Vascular disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes